CLINICAL TRIAL: NCT04593693
Title: A Dual-center Study Evaluating Clinical Acceptance of a NPWT Wound Care System to Expected Standards of Care in Post-acute Patients With a Variety of Wound Types
Brief Title: A Dual-center Study Evaluating Clinical Acceptance of a NPWT Wound Care System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medela AG (Industry)
Collaborators: Joseph M. Still Research Foundation, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GHC1901
Record Dates: First submitted 2020-09-17; First posted 2020-10-20 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Diabetic Foot Ulcer; Pressure Injury; Pressure Ulcer; Surgical Wound; Acute Wound; Traumatic Wound; Dehiscence; Edema
Keywords: Negative Pressure Wound Therapy; Invia Motion
MeSH Terms: conditions — Diabetic Foot; Pressure Ulcer; Surgical Wound; Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Invia Motion Endure NPWT system (Other): Use of Negative Pressure Wound Thearpy
  Interventions: Device: Invia Motion Endure NPWT system

INTERVENTIONS:
Device: Invia Motion Endure NPWT system — lightweight portable single patient use pump, that provides continous or intermittent operation and multiple negative pressure selection options

SUMMARY:
The purpose of this study is to determine if use of the Medela Invia Motion NPWT system supports acceptable progress towards the goal of therapy when treating patients with a variety of wound types during the evaluation period.

DETAILED DESCRIPTION:
The primary objective is to evaluate whether clinical opinion of product performance results in expected wound response and outcomes when using the Medela Invia Motion Endure NPWT system during 4-week study duration.

* Goal of therapy will be defined by the physician according to initial assessment:

Endpoints (dependent on goal of therapy):

* Decrease in wound volume
* Decrease in size of the tunneling area
* Decrease in size of undermining
* Decrease in amount of slough
* Increase in granulation tissue
* Decrease in edema/periwound swelling
* The wound bed is progressing acceptably towards a transition to another treatment modality such as Moist Wound Healing (MWH), surgical closure, or a flap or graft.

**Study endpoint will be determined by physician at the time of enrollment, when the goal of therapy is documented**

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects ≥18 years of age.
* Signed, informed consent by patient or LAR
* Patient is determined to be in need of NPWT for treatment of a diabetic foot ulcer, pressure injuries, and pressure ulcer, surgical wounds, acute/traumatic wounds and dehisced wounds, abscesses, or to prepare the wound bed for grafting or closure and/or to decrease edema
* Patient is comfortable (e.g. not in pain)
* Patient is willing and able to adhere to treatment protocol.

Exclusion Criteria:

* Patient not willing to comply with follow up (f/u) clinic visits
* Subjects with

  * Necrotic tissue with eschar present
  * Untreated osteomyelitis
  * Non-enteric and unexplored fistulas
  * Malignancy in wound
  * Exposed vasculature
  * Exposed nerves
  * Exposed anastomotic site of blood vessels or bypasses
  * Exposed organs
* Subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.
* Patients with concurrent conditions or co-morbidities that in the opinion of the investigator may compromise patient safety or study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
Goal of therapy: Change in wound volume | Up to 4 week study duration
  Wound measurements will be performed each week and length, width and depth of the wound measured during treatment until goal of the therapy is reached
Goal of therapy: Change in size of the tunneling area | Up to 4 week study duration
  Wound measurements will be performed each week and the tunneling of the wound measured during treatment until goal of the therapy is reached
Goal of therapy: Change in size of undermining | Up to 4 week study duration
  Wound measurements will be performed each week and the undermining of the wound measured during treatment until goal of the therapy is reached
Goal of therapy: Change in amount of slough | Up to 4 week study duration
  Wound measurements will be performed each week and the amount of slough measured during treatment until goal of the therapy is reached
Goal of therapy: Change in granulation tissue | Up to 4 week study duration
  Wound measurements will be performed each week and the amount of granulation tissue measured during treatment until goal of the therapy is reached
Goal of therapy: Change in edema/periwound swelling | Up to 4 week study duration
  Wound measurements will be performed each week and the presence of edema determined during treatment until goal of the therapy is reached
Goal of therapy: The wound bed is progressing acceptably towards a transition to another treatment modality such as Moist Wound Healing (MWH), surgical closure, or a flap or graft | Up to 4 week study duration
  Wound measurements will be performed each week and the wound bed visually determined during treatment until goal of the therapy is reached

SECONDARY OUTCOMES:
Evaluate the ease of use from clinicians | Up to 4 week study duration
  A weekly staff satisfaction survey will be obtained from the wound clinic staff members to determine ease of use on a scale from higher to worse score with four values (more satisfied, satisfied, neutral, less satisfied)
Evaluate overall satisfaction from clinicians | Up to 4 week study duration
  A weekly staff satisfaction survey will be obtained from the wound clinic staff members to determine overall satisfaction with the device on a scale from higher to worse score with four values (more satisfied, satisfied, neutral, less satisfied)

OTHER OUTCOMES:
Determine performance satisfaction of dressing components on periwound | Up to 4 week study duration
  A weekly staff satisfaction survey on the ability to maintain dressing seal will be obtained from the wound clinic staff members to determine performance satisfaction of dressing components on periwound on a scale from higher to worse score with four values (more satisfied, satisfied, neutral, less satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Claus Brandigi, MD, Principal Investigator — Joseph M. Still Research Foundation, Inc.
Locations (2):
- United States (2):
  - Joseph M. Still Burn Center and Wound Clinic at Doctors Hospital, Augusta, Georgia
  - JMS Burn Centers, Inc. at Wellstar Cobb Hospital, Austell, Georgia

IPD SHARING:
Plan to Share IPD: No